CLINICAL TRIAL: NCT03412760
Title: Hydrops: Diagnosing & Redefining Outcomes With Precision Study
Acronym: HyDROPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Fetal Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HydropsUCSF; 5K12HD001262 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hydrops Fetalis; Birth Defect; Fetal Anomaly
Keywords: hydrops fetalis; birth defect; fetal anomaly; exome sequencing
MeSH Terms: conditions — Hydrops Fetalis; Congenital Abnormalities | interventions — Exome

STUDY DESIGN:
Intervention Model Description: All cases of unexplained non-immune hydrops fetalis (NIHF) or other birth defects enrolled in the study will be offered exome sequencing (ES) for the affected fetus or neonate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Exome sequencing (Experimental): There is only one arm of this study. All enrolled participants with unexplained NIHF or other birth defect will be offered exome sequencing for the affected fetus or neonate. Please refer to the Study Design section for further details.
  Interventions: Diagnostic Test: Exome sequencing

INTERVENTIONS:
Diagnostic Test: Exome sequencing — Expansive genetic test performed for affected fetus or neonate.

SUMMARY:
This is a national, prospective study designed to investigate the genetic etiologies of non-immune hydrops fetalis (NIHF) and other birth defects. At least half of prenatally diagnosed NIHF cases remain of unknown etiology after standard work up, and a substantial proportion of other birth defects remain of unknown etiology as well. The investigators are performing exome sequencing (ES) for the affected fetus or neonate in unexplained cases, as well as enrolling cases with a genetic explanation to represent the full spectrum of diseases underlying NIHF and other birth defects.

DETAILED DESCRIPTION:
Up to 1:1700 pregnancies are affected by non-immune hydrops fetalis (NIHF), and this condition is associated with significant perinatal risks ranging from preterm birth to Ballantyne (maternal mirror) syndrome, stillbirth, and neonatal death. Birth defects affect 1:33 pregnancies, and are the leading cause of infant death (contributing to approximately 20% of infant deaths). The investigators are performing exome sequencing (ES) for the affected fetus or neonate in unexplained cases, as well as enrolling cases with a genetic explanation to represent the full spectrum of diseases underlying NIHF and other birth defects.

This study is open for enrollment by invitation. In addition to performing ES, the investigators are collecting clinical data prospectively on all cases of NIHF and other birth defects, including demographics, medical and obstetric history, prenatal and delivery course, and postnatal outcomes.

The specific research aims include:

1. Create registry of clinical data for cases of NIHF and other birth defects.
2. Investigate genetic variants underlying NIHF and other birth defects via ES.
3. Characterize the features and outcomes of genetic diseases presenting with NIHF and other birth defects.

   * In particular, the researchers are focused on enrolling cases of increased nuchal translucency, cystic hygroma, abnormal fetal fluid collection (even single fluid compartments such as isolated pleural effusion), and/or frank NIHF.

This research will contribute novel information about the frequency and types of genetic disorders in fetuses and newborns with a diagnosis of NIHF and other birth defects, enabling providers to more accurately counsel about prognosis and individualize perinatal care. This information will also facilitate informed decision-making for parents, allow the care team to anticipate specific perinatal needs, and enable more precise counseling for the parents about recurrence risks for NIHF and other birth defects. Further, the research will facilitate future aims such as novel fetal therapies for genetic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Singletons or dichorionic twin pregnancies that are diagnosed prenatally with non-immune hydrops fetalis (NIHF) or another birth defect. Cases with chromosomal abnormalities, postnatal samples, and stillbirths will still be included.

Exclusion Criteria:

* Monochorionic twin pregnancies and cases of hydrops fetalis that are attributed to red cell alloimmunization (due to hydrops fetalis caused by different pathophysiologic processes).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Genetic variants detected with exome sequencing that implicate a genetic disease underlying non-immune hydrops fetalis (NIHF) and other birth defects. | Turn around time for exome sequencing results is 2-4 weeks for ongoing pregnancies and live infants, and is 8-12 weeks for stillbirths, terminations, and infant demises.
  Both NIHF and birth defects can be caused by a variety of genetic variants that researchers are continuing to learn more about. Exome sequencing will yield information about the specific genetic variants present in cases of NIHF and other birth defects, and about the specific diseases implicated by these variants. Investigators will determine the proportion of cases seen in the setting of particular genetic variants, and will correlate phenotypic outcomes with specific genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Sparks, MD, MAS, Principal Investigator — University of California, San Francisco; Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared only in accordance with NIH/NICHD regulations as the Women's Reproductive Health Research (WRHR) grant is a funding source for this study, and is co-sponsored by these bodies.

REFERENCES:
- [Derived] Sparks TN, Lianoglou BR, Adami RR, Pluym ID, Holliman K, Duffy J, Downum SL, Patel S, Faubel A, Boe NM, Field NT, Murphy A, Laurent LC, Jolley J, Uy C, Slavotinek AM, Devine P, Hodoglugil U, Van Ziffle J, Sanders SJ, MacKenzie TC, Norton ME; University of California Fetal-Maternal Consortium; University of California, San Francisco Center for Maternal-Fetal Precision Medicine. Exome Sequencing for Prenatal Diagnosis in Nonimmune Hydrops Fetalis. N Engl J Med. 2020 Oct 29;383(18):1746-1756. doi: 10.1056/NEJMoa2023643. Epub 2020 Oct 7. PMID 33027564